CLINICAL TRIAL: NCT07356869
Title: Comparative Evaluation of Probiotic-Based Versus Ethyl Lauroyl Arginate-Containing Mouthwashes on Streptococcus Mutans Counts, Dental Plaque Accumulation, and Salivary pH in a Group of Egyptian School Children: A Randomized Controlled Clinical Trial
Brief Title: Probiotic-Based Versus Ethyl Lauroyl Arginate-Containing Mouthwashes on Streptococcus Mutans Counts, Dental Plaque Accumulation, and Salivary pH in a Group of Egyptian School Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Osama Mohamed Abdelrazik, B.D.S, Faculty of Dental Medicine (Cairo-Boys), Al-Azhar University, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1246/4697
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Probiotic; Ethyl Lauroyl Arginate; Mouthwashes; Streptococcus Mutans; Dental Plaque; Salivary pH; Children
MeSH Terms: conditions — Dental Plaque | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Patients will be receive probiotic mouthwash and instructed to rinse 5ml twice daily for 30 seconds for 28 days.
  Interventions: Other: Probiotic mouthwash
- Group B (Experimental): Patients will be treated with ethyl lauroyl arginate-containing mouthwash and instructed to rinse 5ml twice daily for 30 seconds for 28 days.
  Interventions: Other: Ethyl lauroyl arginate mouthwash
- Group C (Active Comparator): Patients will receive professional prophylaxis (scaling + polishing) at baseline and will use only regular toothpaste twice daily, with no adjunctive mouthwashes over 28 days.
  Interventions: Other: Professional prophylaxis (scaling + polishing)

INTERVENTIONS:
Other: Probiotic mouthwash — Patients will be receive probiotic mouthwash and instructed to rinse 5ml twice daily for 30 seconds for 28 days.
  Arms: Group A
Other: Ethyl lauroyl arginate mouthwash — Patients will be treated with ethyl lauroyl arginate mouthwash and instructed to rinse 5ml twice daily for 30 seconds for 28 days.
  Arms: Group B
Other: Professional prophylaxis (scaling + polishing) — Patients will receive professional prophylaxis (scaling + polishing) at baseline and will use only regular toothpaste twice daily, with no adjunctive mouthwashes over 28 days.
  Arms: Group C

SUMMARY:
This study aims to compare the efficacy of probiotic-based mouthwashes versus ethyl lauroyl arginate-containing mouthwashes in reducing Streptococcus mutans count, dental plaque accumulation, and salivary pH among a group of Egyptian schoolchildren.

DETAILED DESCRIPTION:
Dental caries remains one of the most prevalent chronic infectious diseases among Egyptian schoolchildren, with Streptococcus mutans (S. mutans) playing a primary etiological role due to its acidogenic and aciduric properties, which contribute to enamel demineralization and plaque formation.

Ethyl Lauroyl Arginate (LAE), a cationic surfactant derived from lauric acid and arginine, has demonstrated potent bactericidal activity against cariogenic organisms, including S. mutans, while also reducing biofilm formation and preserving oral microbiome balance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Egyptian schoolchildren aged 6-12 years.
* Good general health.
* Mild to moderate dental plaque accumulation.
* Parental/caregiver willingness to provide consent

Exclusion Criteria:

* Antibiotic or antimicrobial use within the last month.
* Allergies to the mouthwash components.
* Systemic diseases affecting oral health.
* Orthodontic appliances or extensive dental restorations.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
S. mutans count | 28 days post-intervention
  S. mutans count will be measured at baseline (0 day) and post-intervention (28 days).

SECONDARY OUTCOMES:
Plaque index score | 28 days post-intervention
  The plaque index score is classified as:
  * Score 0; No plaque
  * Score 1; Mild plaque accumulated along the gingival margin
  * Score 2; Moderate plaques accumulated along the gingival margin
  * Score 3; Heavy plaques accumulated along the gingival margin and adjacent tooth surface.
  Plaque index score will be measured at baseline (0 day) and post-intervention (28 days).
Salivary pH | 28 days post-intervention
  Salivary pH measurements will be carried out by pH strips or pH meter.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University (Faculty of Dentistry), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.